CLINICAL TRIAL: NCT04140513
Title: A Pilot Study to Evaluate the Utility of Interim Digital PET/CT in Predicting Outcomes for Locally Advanced Oropharyngeal Cancer
Brief Title: Digital PET Scan for the Prediction of Outcomes in Patients With Locally Advanced Oropharyngeal Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI decision
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Eric Miller, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OSU-19172; NCI-2019-05315 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2019-10-24; First posted 2019-10-28 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Clinical Stage II HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Clinical Stage III HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Locally Advanced Oropharyngeal Squamous Cell Carcinoma; Pathologic Stage II HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Pathologic Stage III HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Stage III Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage IVA Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage IVB Oropharyngeal (p16-Negative) Carcinoma AJCC v8
MeSH Terms: conditions — Oropharyngeal Neoplasms; Carcinoma | interventions — Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Diagnostic (dPET) (Experimental): Patients receive fludeoxyglucose F-18 via injection and undergo dPET over 20 minutes after standard of care computed tomography (CT) imaging (week -2), after receiving 20-26 Gy and 40-46 Gy of radiation (weeks 3 and 5), and 3 months after completion of treatment. Patients with concern for residual disease may receive an additional dPET 6 months after treatment.
  Interventions: Radiation: Fludeoxyglucose F-18; Procedure: Positron Emission Tomography

INTERVENTIONS:
Radiation: Fludeoxyglucose F-18 — Given via injection
  Other Names: 18FDG; FDG; Fludeoxyglucose (18F); fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Procedure: Positron Emission Tomography — Undergo dPET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This trial studies how well digital PET scan works in predicting outcomes in patients with oropharyngeal cancer that has spread from where it started to nearby tissue or lymph nodes (locally advanced). The development of digital detectors for PET is a technological improvement in medical imaging that could potentially impact many areas of clinical oncology, including staging, radiation planning accuracy, and the assessment of treatment response. Digital technology may improve PET imaging performance by providing better timing, energy and spatial resolution, higher count rate capabilities and linearity, increased contrast, and reduced noise. Utilizing digital PET scan, may work better in predicting outcomes and treatment response in patients with oropharyngeal cancer compared to conventional PET.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the utility of early (i.e. during treatment) digital positron emission tomography (dPET) as a diagnostic tool to predict local control 6 months after definitive chemoradiation for patients with locally advanced oropharyngeal carcinoma.

SECONDARY OBJECTIVES:

I. To study the association between dynamic dPET parameters taken at early time points (i.e. during treatment) and CR on PET after definitive chemoradiation.

II. To study the association between dynamic dPET parameters taken at early time points (i.e. during) treatment and 2 year local control after definitive chemoradiation.

III. To assess the ability of dynamic dPET compared to conventional PET or conventional-equivalent dPET reconstruction to identify tumor volumes with greater sensitivity at the time of before (dPET1), during (dPET2, dPET3) and after (dPET4, dPET5) chemoradiation.

IV. To generate preliminary data for future methodology or clinical trials.

OUTLINE:

Patients receive fludeoxyglucose F-18 via injection and undergo dPET over 20 minutes after standard of care computed tomography (CT) imaging (week -2), after receiving 20-26 Gy and 40-46 Gy of radiation (weeks 3 and 5), and 3 months after completion of treatment. Patients with concern for residual disease may receive an additional dPET 6 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient who will undergo definitive radiation with concurrent chemotherapy with cisplatin 40 mg/m^2 weekly (preferred) or high dose cisplatin 100 mg/m^2 for histologically confirmed locally advanced squamous cell carcinoma of the oropharynx
* Patient must have clinically or radiographically evident measurable disease at the primary site and at nodal station(s). Tonsillectomy or local excision of the primary or nodal disease is not permitted
* p16 and/or human papillomavirus (HPV) status obtained on biopsy specimen (archival or fresh)
* Patients must provide their personal smoking history prior to registration
* Patients must fall into one of the following stage (American Joint Committee on Cancer [AJCC] 8) and risk groups based on pre-treatment work-up and smoking history:

  * Low risk classification:

    * p16 and/or HPV positive, T1-3, N1-2, M0 with =< 10 pack years smoking history OR
  * Intermediate risk classification:

    * p16 and/or HPV positive, T4, N3, M0 and/or HPV positive with > 10 pack year smoking history
    * HPV negative, T1-3, N1-2b, M0, with =< 10 pack years smoking history OR
  * High risk classification:

    * p16 and/or HPV negative, T4, N3, M0
    * p16 and/or HPV negative with > 10 pack year smoking history
* Patients with no contraindications to PET imaging or cisplatin
* No prior history of radiation therapy
* Patient has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Patients with remaining teeth must undergo a dental evaluation prior to enrolment
* Ability to provide informed consent obtained prior to participation in the study and any related procedures being performed
* Women of child-bearing potential (WOCBP) must have a negative pregnancy test within 14 days of the first administration of study treatment. Urine human chorionic gonadotropin (HCG) is an acceptable pregnancy assessment
* Women of child-bearing potential and men who are sexually active should be willing and able to use medically acceptable forms of contraception throughout the treatment phase of the trial and until 60 days following the last study treatment

Exclusion Criteria:

* Prior cancers except non-melanoma skin cancer outside of the head and neck unless disease free for 5 years
* Carcinoma of unknown primary, even if p16 positive
* Clinical or radiologic evidence of metastatic disease as defined by disease below the clavicles
* Simultaneous primary cancers or separate bilateral primary tumor sites with the exception of patients with bilateral tonsil cancers
* Subjects who are breast-feeding, or have a positive pregnancy test will be excluded from the study. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Medical contraindications to PET imaging (e.g. pregnancy, nursing mothers, weight greater than 420 pounds)
* Medical contraindications to cisplatin or prior allergic reaction to cisplatin
* Subjects who are unable to receive intravenous contrast due to a contrast allergy or poor renal function
* Subjects who are prisoners
* Any serious and/or unstable pre-existing medical disorder (aside from malignancy exception above), psychiatric disorder, or other conditions that could interfere with subject?s safety, obtaining informed consent or compliance to the study procedures, in the opinion of the Investigator. This could include severe, active co-morbidities such as:

  * Uncontrolled cardiac disease (hypertension, unstable angina, myocardial infarction within last 6 months, uncontrolled congestive heart failure, cardiomyopathy with decreased ejection fraction)
  * Uncontrolled diabetes
  * Acute bacterial or fungal infection requiring intravenous antibiotics at time of registration
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days of registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10-09 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Quantitative assessments of digital positron emission tomography (dPET) characteristics generated at early time points during treatment | Up to 2 years
  For each of the promising dPET parameters identified in the primary analysis we will examine potential cut-points to be used to best predict 6-month response/non-response using receiver operating characteristic (ROC) methods. Here we will examine specificity, sensitivity, positive predictive value and negative predictive values for each promising parameter to allow for preliminary data to be generated to anticipate which parameters may warrant future study.

SECONDARY OUTCOMES:
Tumor burden | Up to 2 years
  Will compare digital versus conventional PET. Comparison of PET parameters from the dPET or the conventional (c)PET will be visualized using scatterplots; agreement between the two methods will be summarized.
Response rate for each patient local control | At 2 years
  Will be defined as no evidence of disease at 6 months on physical and endoscopic exam for patient with a compete response on 3 month PET. Will be performed using Kaplan-Meier methods.
Progression-free survival (PFS) | Up to 2 years
  PFS will be performed using Kaplan-Meier methods.
Standard uptake volume (SUV) from digital/conventional PET | At 3 months
  Will assess SUV and will compare mean values for each interim dPET. The changes of dPET/cPET SUV over the study period will be visualized using longitudinal plot, summarized at each time point, and modeled using linear mixed model for repeated measures.
Metabolic tumor volume (MTV) from digital/conventional PET | At 3 months
  Will assess MTV and will compare mean values for each interim dPET. The changes of dPET/cPET MTV over the study period will be visualized using longitudinal plot, summarized at each time point, and modeled using linear mixed model for repeated measures.
Total lesion glycolysis (TLG) from digital/conventional PET | At 3 months
  Will calculate TLG based on MTV and SUV and will compare mean values for each interim dPET. The changes of dPET/cPET TLG over the study period will be visualized using longitudinal plot, summarized at each time point, and modeled using linear mixed model for repeated measures.

CONTACTS AND LOCATIONS:
Overall Officials: Eric D Miller, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu